CLINICAL TRIAL: NCT06491329
Title: Effect of Aerobic Interval Training on Atrial Fibrillation Burden：A Multicenter Randomized Controlled Study
Brief Title: Effect of Aerobic Interval Training on Atrial Fibrillation Burden
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZKY-PJ-2024-29
Record Dates: First submitted 2024-06-22; First posted 2024-07-09 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Cardiac Rehabilitation
MeSH Terms: conditions — Atrial Fibrillation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (Experimental): For non-permanent atrial fibrillation patients, a 12-week high-intensity interval training will be administered. The primary objective is to assess alterations in atrial fibrillation burden, with secondary endpoints encompassing changes in cardiorespiratory fitness, quality of life metrics, psychological profiling, atrial strain, ventricular diastolic function, as well as the incidence rates of exercise-related adverse events and adverse cardiovascular events.
  Interventions: Other: high-intensity interval training
- moderate-intensity interval training (Experimental): For non-permanent atrial fibrillation patients, a 12-week moderate-intensity interval training will be administered. The primary objective is to assess alterations in atrial fibrillation burden, with secondary endpoints encompassing changes in cardiorespiratory fitness, quality of life metrics, psychological profiling, atrial strain, ventricular diastolic function, as well as the incidence rates of exercise-related adverse events and adverse cardiovascular events.
  Interventions: Other: moderate-intensity interval training
- Maintain previous exercise habits group (No Intervention): Not undergoing exercise rehabilitation, maintaining previous exercise habits

INTERVENTIONS:
Other: high-intensity interval training — high-intensity interval training ： 40-50 minutes, patients engage in power cycling with intervals of high-intensity exercise at 75%-100% of VO2peak for 30s-1min, followed by 30s-1min of passive recovery, totaling 15-25 cycles.
  Arms: High-intensity interval training
Other: moderate-intensity interval training — 40-50 minutes, involves power cycling with 8 minutes of moderate-intensity exercise at 40%-60% of VO2peak followed by 2 minutes of passive recovery, totaling 4 cycles.
  Arms: moderate-intensity interval training

SUMMARY:
Atrial fibrillation is the most common arrhythmia, with an increasing incidence and prevalence, significantly increasing the risk of death, stroke, heart failure, cognitive impairment, and dementia, severely impacting the quality of life for patients and burdening society and healthcare systems. In recent years, exercise-based cardiac rehabilitation has gradually become a new approach for the treatment of patients with heart disease. The main research topics include: 1. Changes in atrial fibrillation burden in non-permanent atrial fibrillation patients after 12 weeks of HIIT(high-intensity interval training ) or MIIT (moderate-intensity interval training). 2. Changes in cardiorespiratory fitness, quality of life scores, mental health assessment scores, atrial strain, and left ventricular diastolic function in non-permanent atrial fibrillation patients after 12 weeks of aerobic interval training, along with follow-up on the occurrence of exercise-related adverse events and adverse cardiovascular events during the study period.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized clinical trial. It aims to enroll a total of 156 patients with non-permanent atrial fibrillation. Participants will be randomly assigned to the HIIT group, MIIT group, and control group. The HIIT and MIIT groups will receive 12 weeks of high-intensity interval aerobic exercise training and moderate-intensity interval aerobic exercise training, respectively, while the control group will maintain their previous exercise habits.The study will compare the atrial fibrillation burden, cardiorespiratory fitness, quality of life scores, mental health scale scores, blood lipids, blood glucose levels, atrial strain, and ventricular diastolic function changes among patients in the different exercise intervention groups and the control group after 12 weeks. Additionally, the occurrence rates of exercise-related adverse events and cardiovascular adverse events during the follow-up period will be assessed to evaluate the effectiveness and safety of cardiac rehabilitation in the treatment of atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-74 years;
2. Patients with non-permanent atrial fibrillation;
3. Resting heart rate ≤110 beats/min;
4. No history of receiving a formal exercise prescription within the past six months;
5. Willing to participate in this study, provide written informed consent, and agree to comply with follow-up procedures.

Exclusion Criteria:

1. History of myocardial infarction, endocarditis/myocarditis/pericarditis, stroke (ischemic/hemorrhagic), pulmonary embolism, lower extremity venous thrombosis, or cardiac surgery within the past 6 months;
2. Moderate to severe pulmonary arterial hypertension, moderate to severe valvular heart disease, hypertrophic cardiomyopathy, aortic stenosis/dilation/dissection/intramural hematoma, congenital heart disease;
3. Heart failure (NYHA class III-IV) or acute exacerbation of heart failure within the past 3 months;
4. Unstable angina or severe coronary artery disease without revascularization;
5. Concurrent severe arrhythmias

   * frequent multifocal premature ventricular contractions
   * ventricular tachycardia, ventricular fibrillation
   * high-degree or complete atrioventricular block
   * ventricular asystole lasting more than 5 seconds
6. Uncontrolled hypertension or hypotension;
7. Severe renal or hepatic dysfunction

   * Stage 5 chronic kidney disease, defined as glomerular filtration rate <15 ml/(min•1.73 m2) or requiring dialysis;
   * Patient with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than or equal to 5 times the upper limit of normal as defined by the center during screening;
8. Hypoxemia or severe lung disease;
9. Lower extremity arterial stenosis or musculoskeletal disease preventing exercise training;
10. Intracardiac thrombus;
11. Pregnancy;
12. Cognitive impairment preventing study cooperation;
13. Severe anemia, infection, electrolyte disturbances, hyperthyroidism;
14. Planned atrial fibrillation ablation during the study period;
15. Post-implantation of pacemaker or ICD;
16. Inability to use smart devices;
17. Concurrent cancer or autoimmune or systemic inflammatory disease;
18. Regular moderate-to-high intensity exercise habits (≥2 sessions of high-intensity endurance training per week or ≥3 sessions of moderate-intensity endurance training

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation burden | 14 weeks
  The ratio of atrial fibrillation duration to total monitoring time

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 14 weeks
  Peak oxygen consumption (VO2peak)
Severity of atrial fibrillation symptoms | 14 weeks
  Atrial Fibrillation Symptom EHRA Score
General quality of life assessment | 14 weeks
  SF-36 Quality of Life Questionnaire
Prognostic indicators | 14 weeks
  MACE is defined as death, rehospitalization, cardiogenic shock, heart failure, new-onset malignant arrhythmias, stroke, and acute coronary syndrome
Incidence of Exercise-related adverse events (Safety indicators) | 14 weeks
  Exercise-related adverse events are defined as falls during training, muscle ligament strains, headaches/dizziness, vomiting, angina, shortness of breath, syncope, hypotension, new-onset arrhythmias, acute heart failure, acute myocardial ischemia, hypoxemia (oxygen saturation <88%), abnormal elevation or decrease in blood pressure (systolic blood pressure rising to ≥220 mmHg or falling by >20 mmHg or diastolic blood pressure ≥120 mmHg).
Atrial reservoir train | 14 weeks
  the difference of the strain value at the strain curve peak minus end-diastole
Atrial conduit strain | 14 weeks
  the same value as atrial reservoir train, but with a negative sign
Atrial contraction strain | 14 weeks
  the difference of the strain value at end diastole (by definition zero) minus the value at onset of atrial contraction
ventricular diastolic function-1 | 14 weeks
  Interventricular e' velocity
ventricular diastolic function-2 | 14 weeks
  lateral wall e' velocity
Compliance assessment indicators | 14 weeks
  Compliance of the intervention protocol, defined as the total number of actual training sessions completed divided by 36 sessions X 100%; Tolerance of the training protocol, defined as the number of actual training sessions completed according to the planned protocol, intensity, and duration divided by 36 sessions X 100%.
Patient Health Questionnaires Scale | 14 weeks
  PHQ-9 Depression Self-Rating Scale
Gneralized Anxiety Disorder Scale | 14 weeks
  GAD-7 Generalized Anxiety Disorder Scale
Biochemical indicators-1 | 14 weeks
  blood glucose
Biochemical indicators-2 | 14 weeks
  lipids
Biochemical indicators-3 | 14 weeks
  NT-proBNP
Biochemical indicators-4 | 14 weeks
  interleukin
Biochemical indicators-5 | 14 weeks
  C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: YU-TAO GUO, Doctor, Study Chair — Sixth Medical Center of Chinese PLA General Hospital
Locations (1):
- Sixth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott AD, Verdicchio CV, Mahajan R, Middeldorp ME, Gallagher C, Mishima RS, Hendriks JML, Pathak RK, Thomas G, Lau DH, Sanders P. An Exercise and Physical Activity Program in Patients With Atrial Fibrillation: The ACTIVE-AF Randomized Controlled Trial. JACC Clin Electrophysiol. 2023 Apr;9(4):455-465. doi: 10.1016/j.jacep.2022.12.002. Epub 2023 Jan 18. PMID 36752479
- [Background] Reed JL, Terada T, Vidal-Almela S, Tulloch HE, Mistura M, Birnie DH, Wells GA, Nair GM, Hans H, Way KL, Chirico D, O'Neill CD, Pipe AL. Effect of High-Intensity Interval Training in Patients With Atrial Fibrillation: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2239380. doi: 10.1001/jamanetworkopen.2022.39380. PMID 36315143